CLINICAL TRIAL: NCT01583205
Title: Coping Effectiveness Training for Recently Diagnosed ALS Patients and Care Partners
Brief Title: Coping Effectiveness Training for ALS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not funded.
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Judith G. Rabkin, PhD, Research Scientist, Research Foundation for Mental Hygiene, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6514
Record Dates: First submitted 2012-04-05; First posted 2012-04-23 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: ALS; Distress
Keywords: ALS; Coping Effectiveness Training; Distress; Care Giver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coping Effectiveness Training (Experimental): Coping Effectiveness Training -ALS (CET-ALS) is an eight session intervention derived from Coping Effectiveness Training (CET), a manualized intervention based on stress and coping theory. It is designed to strengthen coping skills and alleviate distress for either the patient or care partner following a diagnosis of ALS.
  Interventions: Behavioral: Coping Effectiveness Training - ALS

INTERVENTIONS:
Behavioral: Coping Effectiveness Training - ALS — Eight coping effectiveness training counseling sessions.
  Other Names: CET

SUMMARY:
The investigators propose to adapt and pilot test a behavioral intervention for recently diagnosed patients with Amyotrophic Lateral Sclerosis (ALS), and/or a family care partner. ALS fatal neurodegenerative disease, the diagnosis of which can have a devastating impact on patients and their families. Our eight session intervention is derived from Coping Effectiveness Training, a manualized intervention based on stress and coping theory. It is designed to strengthen coping skills and alleviate distress following diagnosis.

Participants (patients and/or care partners) will be recruited from the Eleanor and Lou Gehrig MDA/ALS Research Center, Columbia University. The main outcomes are changes in distress level, depression and anxiety symptoms, and coping self-efficacy.

Once the investigators gain preliminary experience with the manual, get some sense of feasibility and acceptance, and learn about patient and care partner reactions, the investigators will be better able to prepare a grant application seeking NIH support for the development of the intervention, with the eventual goal of a multisite randomized controlled trial (RCT).

DETAILED DESCRIPTION:
ALS is a rare, devastating, fatal neurodegenerative disease of largely unknown cause. Average survival after diagnosis is about 3 years. The diagnostic process is often protracted, but even though the possibility of ALS may have been mentioned earlier, when the diagnosis is confirmed, patients and family members are often shocked and overwhelmed.

After the diagnostic visit, patients (and accompanying family member) are commonly scheduled to return to the clinic or office in 3 to 6 months. At this first routine clinic visit, the focus is generally on assessment and management of mobility issues, diet, occupational adjustments, advance planning directives, insurance coverage and other pressing issues that usually take up the allotted time. Thus, there is often little opportunity to address the emotional impact of the diagnosis at that visit.

Our goal is a manualized intervention suitable for telephone or Skype delivery, for the management of distress and enhancement of coping skills among recently diagnosed ALS patients and/or their family care partner. We are adapting the intervention developed by Chesney, Folkman and colleagues, "Coping Effectiveness Training," as being the most salient and theoretically powerful design for our purpose. We base our work on Folkman's revised model that incorporates meaning-focused coping and the importance of positive emotions, in addition to the original model of problem-focused and emotion-focused coping. The course of ALS entails progressive losses, of mobility, fine and gross motor skills, speech, swallowing, and respiration. Each requires recalibrating emotional response and coping with new challenges. Early intervention to strengthen coping skills may equip patients and care partners to handle new challenges as they arise, although in this initial study we will not follow patients long enough to observe long-term effects, if present. Based on successful findings in this pilot study, the next step will be to conduct a larger RCT of the intervention.

Specific Aims and Hypotheses

AIM 1. To adapt and refine a manual for Coping Effectiveness Training for recently diagnosed ALS patients and their care partners (CET-ALS) based on Coping Effectiveness Training (CET). We will seek input from interviews with patients (whom we know from their participation in our ongoing studies), care partners and ALS clinic staff.

AIM 2. Feasibility and Acceptability: Evaluate acceptability, attrition, participant satisfaction and perceived barriers and facilitators to intervention delivery.

ELIGIBILITY:
PATIENTS:

Inclusion Criteria:

1. ALS diagnosis (possible, probable, or definite) in the past year
2. Expresses distress (4+) on Distress Thermometer, or symptoms of anxiety or depression (VAS scales)
3. Speaks English
4. Able and willing to give informed consent
5. Speaks clearly enough for telephone communication

Exclusion Criteria:

1. Untreated or under-treated Major Depressive Disorder

CARE PARTNERS:

Inclusion Criteria:

1. Has a family member or close friend diagnosed with ALS (possible, probable, or definite) in the past year
2. Expresses distress (4+) on Distress Thermometer, or symptoms of anxiety or depression (VAS scales)
3. Speaks English
4. Able and willing to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | The PHQ-9 will be given at baseline and then after the particpant completes the 8 counseling sessions (on average ~ 4 months after baseline).
  The Patient Health Questionnaire includes 9 items, each representing one of the 9 diagnostic criteria for major depressive disorder (DSM-IV) plus follow-up probes to ascertain duration, and functional impairment if any. The 4 response options refer to frequency, if present. The scale generates both a numerical score with cut-offs and a diagnostic approximation. It will be clinician-administered, as we have done in other ALS studies, and we will add follow-up queries re: past episodes, if any, as well as ongoing or previous mental health treatment.
Speilberger State Anxiety Inventory (STAI) | The STAI will be given at baseline and then after the particpant completes the 8 counseling sessions (on average ~ 4 months after baseline).
  This 20-item scale assesses current levels of anxiety, excluding somatic symptoms. It is not meant as a diagnostic measure. The response format is a 4-point Likert scale. Items are summed to provide a total severity score. Cut-offs are provided. It has been used successfully in another study of recently diagnosed ALS patients.
Coping Self-Efficacy Scale (13-Item) | The Coping Self-Efficacy Scale will be given at baseline and then after the particpant completes the 8 counseling sessions (on average ~ 4 months after baseline).
  The 26-item scale originally developed by Chesney et al. for CET was subsequently subjected to psychometric analyses using data from 2 randomized trials, and a 13-item version was found to have 3 factors: use of problem-focused coping; stopping unpleasant emotions and thoughts, and getting support from family/friends. The factors showed strong internal consistency reliability and test-retest reliability. The scale is intended to assess a person's ability to cope effectively with life challenges, as well as to assess change in CSE over time in coping-focused intervention research.
Kessler 10-Item Screening Scale for Psychological Distress (K10) | The K10 Scale will be given at baseline and then after the particpant completes the 8 counseling sessions (on average ~ 4 months after baseline).
  The K10 is a quick 10-item screen that is used to assess distress and is shown to be a sensitive screen for DSM-IV anxiety and depressive disorders. The response format is a 5-point Likert scale. Items are summed to provide a total severity score.

CONTACTS AND LOCATIONS:
Overall Officials: Martin C McElhiney, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, Columbia University Medical Center, New York, New York, United States